CLINICAL TRIAL: NCT03123224
Title: Combined Online Assistance for Caregiver Health (COACH): The Efficacy of a Combined Physical Activity and Coping Skills Training Intervention for Caregivers
Brief Title: The COACH Project: Combined Online Assistance for Caregiver Health
Acronym: COACH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Kaci Fairchild, PhD, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAI0003AGG; W81XWH-15-1-0246 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2017-04-03; First posted 2017-04-21 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Traumas, Brain; Alzheimer Disease; Dementia; Head Injury; Concussion, Brain; TBI
Keywords: Caregiver; Caregiving; TBI; dementia; Alzheimer's disease; physical exercise; physical activity; psychosocial; caregiver skills training
MeSH Terms: conditions — Brain Injuries, Traumatic; Alzheimer Disease; Dementia; Craniocerebral Trauma; Brain Concussion; Motor Activity | interventions — Pliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined Aerobic and Resistance Exercise (Experimental): Participants will work with study staff to develop an individualized physical training program based on their level of functioning at study entry. Exercises will focus on increasing the heart rate to a point at which participants will breathe more heavily and may sweat.
  Interventions: Behavioral: Combined Aerobic and Resistance Exercise + Caregiver Skills Training
- Balance and Flexibility (Active Comparator): Participants will work with study staff to develop an individualized physical training program based on their level of functioning at study entry.
  Interventions: Behavioral: Stretching Balance and Flexibility + Caregiver Skills Training

INTERVENTIONS:
Behavioral: Combined Aerobic and Resistance Exercise + Caregiver Skills Training — The combined moderate to high intensity combined aerobic and resistance exercise training + skills training group consists of six months of physical exercise + caregiver skills training followed by an additional six months of follow-up for a total study duration of twelve months. All aspects of these combined interventions will be delivered through mobile technology thus obviating some of the obstacles to caregivers face in meeting their own needs. Caregivers will be provided with study issued equipment (e.g., exercise equipment, activity monitoring devices, and tablets) to complete all elements of the intervention.
  Arms: Combined Aerobic and Resistance Exercise
Behavioral: Stretching Balance and Flexibility + Caregiver Skills Training — The stretching, balance and flexibility training + skills training group consists of six months of physical exercise + caregiver skills training followed by an additional six months of follow-up for a total study duration of twelve months. All aspects of these combined interventions will be delivered through mobile technology thus obviating some of the obstacles to caregivers face in meeting their own needs. Caregivers will be provided with study issued equipment (e.g., exercise equipment, activity monitoring devices, and tablets) to complete all elements of the intervention.
  Arms: Balance and Flexibility

SUMMARY:
This study evaluates the effect of a physical exercise + caregiver skills training on feelings of burden, mood, and biological markers of inflammation in persons who provide care for Veterans with a TBI or dementia. Half of the caregivers will participate in a balance and flexibility + caregiver skills training program, while the other half will participate in a moderate/high intensity aerobic and resistance + caregiver skills training program.

ELIGIBILITY:
Inclusion Criteria:

1. individuals aged 18 - 85
2. distress associated with being the primary caregiver of a person with TBI or dementia
3. endorsement of at least two of the following items: felt overwhelmed, felt like needed to cry, angry or frustrated, distant or cut of from family or friends, moderate to high levels of stress, felt their health had declined
4. provide at least one hour of care (supervision or direct assistance) per week over the past three months
5. approval by Primary Care Provider to participate in physical exercise
6. be proficient in spoken and written English

Exclusion Criteria:

1. current or lifetime history of any psychiatric disorder with psychotic features
2. prominent suicidal or homicidal ideation
3. current alcohol or substance abuse
4. diagnosis of probable or possible dementia
5. a Short Portable Mental Status score of ≥ 8
6. participation in another caregiver intervention within the past year
7. lack of regular access to the internet
8. planned transfer of care recipient to another caregiver or nursing home within 12 months; 8) current severe cardiac disease (e.g., uncontrolled atrial fibrillation, defined as mean 24 hour heart rate >85 beats/min, or 24 hour maximal ventricular rate >150 beats/min; uncontrolled ventricular arrhythmias, defined as recurrent ventricular tachycardia >3 beats in succession, or 24 hour PVC count >20%; active pericarditis or myocarditis; Class III/IV heart failure and / or ejection fraction < 20%; thrombophlebitis; pulmonary disease with a drop in O2 Sat with exercise to 90% without oxygen; embolism within past 6 months)
9. inability to participate in an exercise stress test
10. morbid obesity (BMI > 39)
11. inability to read, verbalize understanding and voluntarily sign the Informed Consent.

Caregivers meeting any of these exclusion criteria will be excluded from all aspects of this project.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden using Zarit Burden Inventory | Six Months
  Zarit Burden Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No